CLINICAL TRIAL: NCT05749965
Title: Unicompartimental Knee Arthroplasties When Borders Are Crossed : Survival Study at 7 Years
Brief Title: Results of Unicompartmental Knee Arthroplasties in Patients Beyond Historical Indications (PUCIL)
Acronym: PUCIL
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, FERNANDEZ Andrea, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2022PI091
Record Dates: First submitted 2023-02-08; First posted 2023-03-01 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Knee Disease
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Limit indications: Obèse (BMI>30), ACL déficiency, HKA > 10°, flessum >10° [HKA : hop knee angle]
  Interventions: Procedure: Unicompartmental knee arthroplasty
- Historical indications: Patient with a BMI between 18,5 and 30, HKA <10°, functionnal ACL, no flessum or <5°
  Interventions: Procedure: Unicompartmental knee arthroplasty

INTERVENTIONS:
Procedure: Unicompartmental knee arthroplasty — medial unicompartmental knee arthroplasty

SUMMARY:
Primary objective:

To compare medial uni compartimental knee arthroplasty between patients who had a limit factor prior to the surgery ans patients who fill thé historical criteria.

Secondary objectives

1 to compare survival of medial UKA between patients with one limit factor and those with multiple limits.

2. To identify the prognosis factors of failure in medial UKA in our center during the time of our analysis (2009-2015)

DETAILED DESCRIPTION:
7 year follow up survival if no amputation or no removal of UKA for TKA

ELIGIBILITY:
Inclusion Criteria:

- medial UKA implanted between 2009 and 2015 at the CCEG

Exclusion Criteria:

* no other UKA
* lost to follow up
* patient refuses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All medial UKA implanted between 2009 and 2015 at the CCEG with follow up at 7 years
Sampling Method: Non-Probability Sample
Enrollment: 522 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Survival of medial UKA | 7 years
  UKA changed or replaced by TKA

SECONDARY OUTCOMES:
to compare UKA survival if multiple limit indication | 7 years
  UKA changed or replaced by TKA
to identify prognostic factors of re operation of patients with a medial UKA implanted between 2009 and 2015 at the CCEG | 7 years
  ACL, flessum, HKA, weight

CONTACTS AND LOCATIONS:
Overall Officials: Andre Fernandez, Study Director — Central Hospital, Nancy, France
Locations (1):
- Centre Chirurgical Emile Gallé, Nancy, France

IPD SHARING:
Plan to Share IPD: No